CLINICAL TRIAL: NCT01182155
Title: Breath Analysis for Evaluation of Radiation Exposure in Lung Cancer Patients Treated With Radiation: A Feasibility Study
Brief Title: Breath Analysis for Evaluation of Radiation Exposure in Lung Cancer Patients Treated With Radiation
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: LUN0043; SU-08102010-6705 (Other: Stanford University)
Record Dates: First submitted 2010-08-12; First posted 2010-08-16 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: Lung Cancer Non-Small Cell Cancer (NSCLC); Lung Cancer Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Exhaled Breath Sampling — Standard of care
  Other Names: breath gas analysis

SUMMARY:
Patients treated with radiation therapy for lung tumors can experience inflammation after treatment. This study hopes to evaluate the use of breath analysis to evaluate changes in the composition of exhaled breath in patients undergoing radiotherapy. If changes can be detected, this may ultimately serve as biomarkers for identifying patients at highest risk for radiation-induced lung injury (radiation pneumonitis).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any type of lung tumor
* Medical recommendation (independent of the study) that the patient undergo thoracic radiation therapy. Radiation therapy may be either fractionated or hypofractionated (i.e. radiosurgery)
* Age >= 18 years old
* Any gender and any ethnic background will be recruited
* Capable of giving written informed consent

Exclusion Criteria:

* Inability of giving written informed consent
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung tumors who are undergoing radiation therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pre and post-radiation FeNO (fraction of exhaled nitric oxide) measurements | Every 3 months for 1 year

SECONDARY OUTCOMES:
Pre and post-radiation CO (carbon monoxide), CO2 (carbon dioxide), and N2O (nitrous oxide) measurements and feasibility as the fraction of patients unable to give a breath sample. Adverse events are not expected but any that appear related to the breath | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Maximilian Diehn MD/PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States